CLINICAL TRIAL: NCT01337739
Title: Use of Dexmedetomidine for Deep Sedation in Patients Undergoing Outpatient Hysteroscopic Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study drug delayed time of discharge which is clinically impracticable.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Shireen Ahmad, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00027663
Record Dates: First submitted 2010-04-19; First posted 2011-04-19 (Estimated); Results first posted 2013-07-12 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-05

CONDITIONS: Pain
Keywords: Hysteroscopic Surgery; Dexmedetomidine; Sedation; Opioids
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Comparator (Placebo Comparator): Continuous infusion of placebo during operative procedure
  Interventions: Drug: Placebo Comparator
- Active Comparator (Active Comparator): Administration of Dexmedetomidine
  Interventions: Drug: Active Comparator

INTERVENTIONS:
Drug: Placebo Comparator — Placebo administration (.9 normal saline sterile)
  Arms: Placebo Comparator
Drug: Active Comparator — Administration of Dexmedetomidine
  Arms: Active Comparator

SUMMARY:
Patients undergoing deep sedation for outpatient procedures typically receive a combination of benzodiazepines, propofol, and opioids. Side effects of such anesthetics include respiratory depression, nausea and vomiting, and urinary retention, with resultant extended hospital stays and unanticipated admission. The use of dexmedetomidine for deep sedation may increase patient safety by maintaining respiratory drive, while providing sedation, hypnosis, and analgesia. Furthermore, patients may experience decreased pain, nausea, and time to discharge in the PACU, especially if dexmedetomidine decreases the requirement of other drugs such as opioids.

The hypothesis of this study is administration of dexmedetomidine during deep sedation for ambulatory hysteroscopic surgery will result in a 50% reduction of intraoperative opioid compared to sedation with propofol.

DETAILED DESCRIPTION:
Patients will be recruited up to 21 days prior to the day of surgery. Preoperatively: A full preoperative assessment will be completed. Preoperatively, patients will be instructed on the proper use of the verbal rating scale (VRS) for pain and nausea scores. Patients will be randomized by a computer-generated scheme to receive prepared infusions containing either dexmedetomidine (4grams per milliliter or propofol (10 milligrams per milliliter) intraoperatively. The study drug infusions will be prepared by study personnel who are not involved in the assessments. Patients, medical personnel other than the anesthesiologist, and outcome assessors will be blinded to treatment allocation. Only the anesthesiologist administering the treatment infusion and medications intraoperatively will be aware of group allocation.

Intraoperatively: A standardized intraoperative anesthetic plan will be utilized by the anesthesia personnel.All patients will receive premedication with midazolam 2 milligrams intravenous bolus and ketorolac 30 milligrams via the intravenous catheter.

Intraoperative monitoring will include standard monitoring which includes noninvasive blood pressure, electrocardiography, pulse oximetry, and capnography. In addition transcutaneous CO2 will be monitored using the Tosca monitor.(Radiometer, Basel, Austria).

The study drug infusion will be started as either dexmedetomidine (1gram per kilogram over 10 min as a loading dose, followed by a maintenance infusion 0.2 to 1.5 grams per kilogram or propofol (started at 75gram per kilogram per minute and ranging from 12.5 to 125 gram per kilogram per minute titrated to maintain the Observer's Assessment of Alertness/Sedation Scale (OAA/SS) between 0-1. Intraoperative fluids will be restricted to 500 milliliter + 100mililiterml of Lactated Ringer's solution. At the onset of the procedure, the anesthesiologist will administer 0.7gram/kilogram bolus of fentanyl intravenous, followed by additional 25-50gram boluses for any patient movement to surgical stimulus. All patients will receive ondansetron 4 milligram IV 15-20 minutes prior to the end of surgery. Patients will receive glycopyrrolate 0.2 mg IV if HR decreases below 50 bpm.

Postoperatively:

In the recovery room, VRS for pain will be assessed upon admission and at 30 minute intervals thereafter. Analgesics will be administered according to the severity of the pain and degree of alertness.Vomiting and retching episodes.will be assessed at 30 minute intervals using a VRS, and patients with scores greater than 4 or those who request antiemetic treatment will be treated with metoclopramide 10 mg IV.

Recovery from anesthesia and return of psychomotor ability will be assessed using the Modified Post Anesthesia Discharge Scoring System (MPADSS). A score of 8 or greater will indicate discharge readiness. Discharge readiness requires that a patient be awake and alert with stable vital signs, able to ambulate without assistance, and free of side effects. 24 hours after discharge.

Times from end of surgery to oral intake and readiness for discharge, , and all adverse events and medications administered will be recorded. These data will be recorded by research staff blinded to the study group assignments. Subjects will be contacted by telephone 24 hours after surgery to obtain post-discharge data, including a repeat QoR-40 assessment.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Age: 18-64 years
* Female
* Surgery: Gynecologic hysteroscopy
* Language: English speaking
* Consent: Obtained

Exclusion Criteria:

* Pregnant or breast feeding
* Significant arrhythmia or high degree atrioventricular nodal block
* Significant hepatic or renal dysfunction
* Chronic use or addiction to opiates or sedatives
* History of heavy alcohol usage (>4 drinks/day)
* Psychiatric or emotional disorder
* Chronic use of α2-agonists
* Patients with OSA or BMI greater than 30
* Allergy to study drug or anesthetic medications utilized in the protocol

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2010-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shireen Ahmad, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Prentice Womens Hospital, Chicago, Illinois

REFERENCES:
- [Background] Bhananker SM, Posner KL, Cheney FW, Caplan RA, Lee LA, Domino KB. Injury and liability associated with monitored anesthesia care: a closed claims analysis. Anesthesiology. 2006 Feb;104(2):228-34. doi: 10.1097/00000542-200602000-00005. PMID 16436839
- [Background] Panzer O, Moitra V, Sladen RN. Pharmacology of sedative-analgesic agents: dexmedetomidine, remifentanil, ketamine, volatile anesthetics, and the role of peripheral mu antagonists. Crit Care Clin. 2009 Jul;25(3):451-69, vii. doi: 10.1016/j.ccc.2009.04.004. PMID 19576524
- [Background] Bhana N, Goa KL, McClellan KJ. Dexmedetomidine. Drugs. 2000 Feb;59(2):263-8; discussion 269-70. doi: 10.2165/00003495-200059020-00012. PMID 10730549
- [Background] Kaygusuz K, Gokce G, Gursoy S, Ayan S, Mimaroglu C, Gultekin Y. A comparison of sedation with dexmedetomidine or propofol during shockwave lithotripsy: a randomized controlled trial. Anesth Analg. 2008 Jan;106(1):114-9, table of contents. doi: 10.1213/01.ane.0000296453.75494.64. PMID 18165564
- [Background] Taghinia AH, Shapiro FE, Slavin SA. Dexmedetomidine in aesthetic facial surgery: improving anesthetic safety and efficacy. Plast Reconstr Surg. 2008 Jan;121(1):269-276. doi: 10.1097/01.prs.0000293867.05857.90. PMID 18176230
- [Background] Koroglu A, Teksan H, Sagir O, Yucel A, Toprak HI, Ersoy OM. A comparison of the sedative, hemodynamic, and respiratory effects of dexmedetomidine and propofol in children undergoing magnetic resonance imaging. Anesth Analg. 2006 Jul;103(1):63-7, table of contents. doi: 10.1213/01.ANE.0000219592.82598.AA. PMID 16790627
- [Background] Bergese SD, Khabiri B, Roberts WD, Howie MB, McSweeney TD, Gerhardt MA. Dexmedetomidine for conscious sedation in difficult awake fiberoptic intubation cases. J Clin Anesth. 2007 Mar;19(2):141-4. doi: 10.1016/j.jclinane.2006.07.005. PMID 17379129
- [Background] McCutcheon CA, Orme RM, Scott DA, Davies MJ, McGlade DP. A comparison of dexmedetomidine versus conventional therapy for sedation and hemodynamic control during carotid endarterectomy performed under regional anesthesia. Anesth Analg. 2006 Mar;102(3):668-75. doi: 10.1213/01.ane.0000197777.62397.d5. PMID 16492813
- [Background] Arain SR, Ebert TJ. The efficacy, side effects, and recovery characteristics of dexmedetomidine versus propofol when used for intraoperative sedation. Anesth Analg. 2002 Aug;95(2):461-6, table of contents. doi: 10.1097/00000539-200208000-00042. PMID 12145072
- [Background] Tufanogullari B, White PF, Peixoto MP, Kianpour D, Lacour T, Griffin J, Skrivanek G, Macaluso A, Shah M, Provost DA. Dexmedetomidine infusion during laparoscopic bariatric surgery: the effect on recovery outcome variables. Anesth Analg. 2008 Jun;106(6):1741-8. doi: 10.1213/ane.0b013e318172c47c. PMID 18499604
- [Background] Chernik DA, Gillings D, Laine H, Hendler J, Silver JM, Davidson AB, Schwam EM, Siegel JL. Validity and reliability of the Observer's Assessment of Alertness/Sedation Scale: study with intravenous midazolam. J Clin Psychopharmacol. 1990 Aug;10(4):244-51. PMID 2286697
- [Background] Chung F. Discharge criteria--a new trend. Can J Anaesth. 1995 Nov;42(11):1056-8. doi: 10.1007/BF03011083. PMID 8590498

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were introduced to the study in a clinic setting and allowed to review the consent prior to their operative procedure.
Pre-assignment Details: 10 subjects were approached and all of the subjects agreed to participate.
Period: Overall Study
Arm/Group | Placebo Comparator | Active Comparator
Started | 6 | 4
Completed | 6 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All 10 subjects participating were used in final analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Comparator | Active Comparator | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 10
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 43.6 (8.4) | 41.5 (7.43) | 42.8 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Will be the Difference in Intraoperative Opioid (Fentanyl) Administration Between Patients Receiving Dexmedetomidine and Those Receiving Propofol.
Description: The primary outcome will be the difference in intraoperative opioid (fentanyl) administration between patients receiving dexmedetomidine and those receiving propofol. As described by mean and standard deviation.
Time Frame: Interoperative period
Measure: Mean (Standard Deviation); unit: Total Morphine Equivalents mg
Arm/Group | Placebo Comparator | Active Comparator
Number analyzed (Participants) | 6 | 4
Total Morphine Equivalents mg | 11.8 (3.5) | 11.58 (4.79)

2. Secondary Outcome: Time to Discharge
Description: Time to discharge from the Post Anesthesia Care Unit or home or to hospital room.
Time Frame: 24 Hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo Comparator | Active Comparator
Number analyzed (Participants) | 6 | 4
minutes | 88.16 (30) | 115 (33.7)

ADVERSE EVENTS:
Arm/Group | Placebo Comparator | Active Comparator
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 0/6 | 0/4

LIMITATIONS AND CAVEATS:
Early termination of the study due to increased discharge time from the post anesthesia care unit with subjects receiving dexmedetomidine. The delay was consistent among the group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No